CLINICAL TRIAL: NCT03364608
Title: A Randomized, Double-blind, Single Dose, Placebo-controlled, 5-Period, 5-Treatment, Crossover, Multi-center, Dose-ranging Study to Compare PT007 to Placebo MDI and Open-Label Proventil® HFA in Adult and Adolescent Subjects With Mild to Moderate Asthma (ANTORA)
Brief Title: Study to Compare PT007 to Placebo MDI and Open-Label Proventil® HFA in Adult and Adolescent Subjects With Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D6930C00001
Record Dates: First submitted 2017-12-01; First posted 2017-12-06 (Actual); Results first posted 2019-07-24 (Actual); Last update posted 2019-07-24 (Actual); Status verified 2019-07

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Albuterol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- • AS MDI 90 µg (Experimental): (2 actuations of 45 µg/actuation)
  Interventions: Drug: AS MDI 90 μg
- • AS MDI 180 µg (Experimental): (2 actuations of 90 µg/actuation)
  Interventions: Drug: AS MDI 180 µg
- • Placebo MDI (Placebo Comparator): (2 actuations)
  Interventions: Other: Placebo MDI
- • Proventil 90 µg (Active Comparator): (1 actuation of 90 µg/actuation)
  Interventions: Drug: Proventil 90 μg
- • Proventil 180 µg (Active Comparator): (2 actuations of 90 µg/actuation)
  Interventions: Drug: Proventil 180 μg

INTERVENTIONS:
Drug: AS MDI 90 μg — AS MDI 90 μg (2 actuations of 45 μg/actuation)
  Other Names: AS MDI
  Arms: • AS MDI 90 µg
Drug: AS MDI 180 µg — AS MDI 180 μg (2 actuations of 90 μg/actuation)
  Other Names: AS MDI
  Arms: • AS MDI 180 µg
Other: Placebo MDI — Placebo MDI (2 actuations)
  Arms: • Placebo MDI
Drug: Proventil 90 μg — Proventil 90 μg (1 actuation of 90 μg/actuation)
  Other Names: Proventil
  Arms: • Proventil 90 µg
Drug: Proventil 180 μg — Proventil 180 μg (2 actuations of 90 μg/actuation)
  Other Names: Proventil
  Arms: • Proventil 180 µg

SUMMARY:
This is a randomized, double-blind, single-dose, placebo-controlled, 5-period, 5-treatment, crossover, multi-center study to assess the bronchodilatory effect and safety of 2 dose levels of Albuterol Sulfate Pressurized Inhalation Suspension (hereafter referred to as AS MDI), 90 μg and 180 μg, compared with placebo for AS MDI (hereafter referred to as Placebo MDI) and open-label Proventil® hydrofluoroalkane (HFA; hereafter referred to as Proventil) 90 μg and 180 μg in adult and adolescent subjects with mild to moderate asthma. This study design utilizes 10 treatment sequences.

DETAILED DESCRIPTION:
This is a 5-period crossover study. Each Treatment Period is 1 day. Subjects will receive a single dose of randomized study drug at each of the 5 Treatment Visits (Visits 2, 3, 4, 5, and 6), with a 3- to 7-day Washout Period between Treatment Visits.

ELIGIBILITY:
Inclusion Criteria

* Are at least 12 years of age and no older than 65 years
* Have stable (for 6 months) physician-diagnosed asthma with historical documentation of the diagnosis
* Must be receiving 1 of the following required inhaled asthma therapies listed below for at least the last 30 days; Only SABA, which is used as needed for rescue, or Low to medium doses of ICS (alone or in combination with LABA), used regularly as maintenance asthma therapy
* Demonstrate acceptable spirometry performance (ie, meet American Thoracic Society [ATS]/European Respiratory Society [ERS] acceptability/repeatability criteria
* Pre-bronchodilator FEV1 of ≥40 to <90% predicted normal value after withholding SABA for ≥6 hours
* Confirmed FEV1 reversibility to Ventolin, defined as a post-Ventolin increase in FEV1 of ≥15%
* only 2 reversibility testing attempts are allowed

Exclusion Criteria:

* Chronic obstructive pulmonary disease or other significant lung disease (eg, chronic bronchitis, emphysema, bronchiectasis with the need of treatment, cystic fibrosis, or bronchopulmonary dysplasia)
* Oral corticosteroid use (any dose) within 6 weeks
* Current smokers, former smokers with >10 pack-years history, or former smokers who stopped smoking <6 months (including all forms of tobacco, e-cigarettes [vaping], and marijuana)
* Life-threatening asthma as defined as any history of significant asthma episode(s) requiring intubation associated with hypercapnia, respiratory arrest, hypoxic seizures, or asthma-related syncopal episode(s)
* Historical or current evidence of a clinically significant disease
* Cancer not in complete remission for at least 5 years
* Hospitalized for psychiatric disorder or attempted suicide within 1 year
* Unable to abstain from protocol-defined prohibited medications during the study

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-12-15 (Actual); Primary Completion 2018-03-30 (Actual); Study Completion 2018-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Research Site, Rolling Hills Estates, California
  - Research Site, Stockton, California
  - Research Site, Winter Park, Florida
  - Research Site, North Dartmouth, Massachusetts
  - Research Site, St Louis, Missouri
  - Research Site, Raleigh, North Carolina
  - Research Site, Cincinnati, Ohio
  - Research Site, Medford, Oregon
  - Research Site, Spartanburg, South Carolina
  - Research Site, El Paso, Texas

REFERENCES:
- [Derived] Cappelletti C, Maes A, Rossman K, Gillen M, LaForce C, Kerwin EM, Reisner C. Dose-Ranging and Cumulative Dose Studies of Albuterol Sulfate MDI in Co-Suspension Delivery Technology (AS MDI; PT007) in Patients with Asthma: the ASPEN and ANTORA Trials. Clin Drug Investig. 2021 Jun;41(6):579-590. doi: 10.1007/s40261-021-01040-7. Epub 2021 Jun 4. PMID 34089147
- See also: Protocol — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14724&filename=PT007001_Protocol_Redacted_PDFA.pdf
- See also: Statistical Analysis Plan (SAP) — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=14724&filename=PT007001_SAP_Redacted_PDFA.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 sites in the United States, from December 2017 to March 2018. The study was anticipated to run for at least 23 days but not to exceed 68 days.
Pre-assignment Details: Subjects were randomized into one of 10 treatment sequences. Each sequence comprised all 5 treatments included in this study (ie, AS MDI 90 μg, AS MDI 180 μg, Placebo MDI, Proventil 90 μg, and Proventil 180 μg) in a randomized order
Groups:
- Subjects: ITT Analysis set
Period: Overall Study
Arm/Group | Subjects
Started (ITT Analysis Set) | 86
Placebo MDI ((2 actuations)) | 82
AS MDI 90 µg ((2 actuations of 45 µg/actuation)) | 81
AS MDI 180 µg ((2 actuations of 90 µg/actuation)) | 81
Proventil 90 µg ((1 actuation of 90 µg/actuation)) | 82
Proventil 180 µg ((2 actuations of 90 µg/actuation)) | 79
Completed | 78
Not Completed | 8
Not completed — Withdrawal by Subject | 4
Not completed — Protocol Violation | 2
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Population: Overall number of Baseline Participants is from the Safety set.
Groups:
- Overall Study: Safety Set
Arm/Group | Overall Study
Number analyzed (Participants) | 86
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: Safety Set
  Years | 42.7 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Safety Set
  Participants
    Female | 47
    Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Set
  Participants
    Hispanic or Latino | 14
    Not Hispanic or Latino | 72
    Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Safety Set
  Participants
    American Indian or Alaska Native | 0
    Asian | 1
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 20
    White | 62
    More than one race | 0
    Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in FEV1 AUC0-6
Description: Change from baseline in FEV1 (Forced expiratory volume in 1 second) AUC0-6 (Area under the curve from 0 to 6 hours) (spirometry will be obtained at 5, 15, 30, 45, 60, 120, 180, 240, 300, and 360 minutes post-dose) normalized for length of follow up.
Time Frame: Over 6 hours post dose on Day 1
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Groups:
- AS MDI 180 µg; Proventil 180 µg: (2 actuations of 90 µg/actuation)
- AS MDI 90 µg: (2 actuations of 45 µg/actuation)
- Proventil 90 µg: (1 actuation of 90 µg/actuation)
- Placebo MDI: (2 actuations)
Arm/Group | AS MDI 180 µg | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg | Placebo MDI
Number analyzed (Participants) | 79 | 79 | 77 | 78 | 78
Liters | 0.266 [0.219 to 0.313] | 0.203 [0.156 to 0.251] | 0.282 [0.234 to 0.329] | 0.240 [0.193 to 0.288] | 0.070 [0.022 to 0.117]

2. Secondary Outcome: Change From Baseline in FEV1 AUC0-4
Description: Change from baseline in FEV1 (Forced expiratory volume in 1 second) AUC0-4 (Area under the curve from 0 to 4 hours) (spirometry will be obtained at 5, 15, 30, 45, 60, 120, 180, and 240 minutes post-dose) normalized for length of follow up.
Time Frame: Over 4 hours post dose on Day 1
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AS MDI 180 µg | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg | Placebo MDI
Number analyzed (Participants) | 79 | 79 | 77 | 78 | 78
Liters | 0.331 [0.280 to 0.381] | 0.263 [0.213 to 0.313] | 0.349 [0.299 to 0.400] | 0.297 [0.247 to 0.348] | 0.080 [0.030 to 0.131]

3. Secondary Outcome: Peak Change From Baseline in FEV1
Description: Peak Change from baseline in FEV1 (Forced expiratory volume in 1 second)
Time Frame: Over 6 hours post dose on Day 1
Population: mITT Population
Measure: Least Squares Mean (95% Confidence Interval); unit: Liters
Arm/Group | AS MDI 180 µg | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg | Placebo MDI
Number analyzed (Participants) | 79 | 79 | 77 | 78 | 78
Liters | 0.509 [0.451 to 0.567] | 0.433 [0.375 to 0.491] | 0.516 [0.458 to 0.574] | 0.472 [0.414 to 0.530] | 0.233 [0.176 to 0.291]

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time the subject signed informed consent throughout the treatment period and up to 14 days following the last dose of study drug
Description: Serious Adverse Events were collected from the time the subject signed informed consent throughout the treatment period and up to approximately 68 days, which includes screening and follow up (3-7 days after last dose of study drug).
Arm/Group | Placebo MDI | AS MDI 90 µg | Proventil 180 µg | Proventil 90 µg | • Proventil 180 µg
All-Cause Mortality (participants affected / at risk) | 0/82 | 0/81 | 0/81 | 0/82 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81 | 0/81 | 0/82 | 0/79
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81 | 0/81 | 0/82 | 0/79

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Drafts of any and all publications or presentations of this study must be submitted at least 30 days prior to submission for publication or presentation to Pearl Therapeutics for review, approval, and to ensure consistency. Pearl Therapeutics has the right to request appropriate modification to correct facts and to represent it's opinions, or the opinions of the publication committee, if these differ with the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/08/NCT03364608/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03364608/SAP_001.pdf